CLINICAL TRIAL: NCT04787068
Title: Providing Support to Caregivers of Frail Older Adults With Cognitive Impairments
Brief Title: Support for Caregivers of Older Adults With Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Ralph C. Wilson Jr. Foundation (Funding source) (Unknown)
Responsible Party: Principal Investigator, Machiko R Tomita, Clinical Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001647
Record Dates: First submitted 2020-02-25; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Caregiver Burden; Depression; Confidence, Self; Cognition; Fatigue; Function
Keywords: Informal caregivers; Intervention
MeSH Terms: conditions — Caregiver Burden; Depression; Fatigue

STUDY DESIGN:
Intervention Model Description: Experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Intervention is occupational therapy support
  Interventions: Behavioral: Occupational Therapy support
- Control group (No Intervention): No intervention was provided, only educational material was given.

INTERVENTIONS:
Behavioral: Occupational Therapy support — Intervention include (a) didactic education about diseases; (b) the use of errorless techniques to improve assistance for CR's Activities of Daily Living (ADL), Instrumental ADL, and communication tasks; (c) the use of incentives (e.g., providing a favorite scented shampoo); (e) use of a schedule/calendar on a computer, cell phone and/or blackboard in CR's home to coordinate caregiving tasks for family members; (f) suggesting more frequent PACE daycare visits or use of a nearby PACE, having a snack or short game to prevent going to bed right after dinner); (d) use of the Buffalo Functional Exercise for strengthening ( a home-based exercise developed for PACE by the PI and shown to be effective in preventing falls)
  Arms: Treatment group

SUMMARY:
This randomized control study is to test effectiveness of occupational therapy support for informal caregivers of older adults with cognitive decline. Care recipients are community-living older adults who are eligible for a nursing home level of care. At baseline challenges that caregivers are facing will be expressed and individualized solutions will be identified and delivered for the treatment and educational material will be given to the control group. Two and four months later, follow up interview will be made to identify changes in burden, depression, fatigue, self-efficacy, and positive aspect of care giving. It is expected to show when the effectiveness becomes clear.

DETAILED DESCRIPTION:
Family caregivers of frail older adults with cognitive impairments face special challenges in caring for their care recipients (CR) due to their fast declining health. Examples of difficulties include managing CR's behaviors and daily activities, as well as maintaining their own psychological and physical health, which result in high caregiver burden. The aim is to support these caregivers of older adults who are enrollees of the Program for All-inclusive Care for the Elderly (PACE) through occupational therapy (OT) interventions to reduce caregiver burden and depression, and increase positive aspects of caregiving and self-efficacy. Since PACE organizations offer limited support for caregivers due to understanding, supervised OT graduate students (OTGS) will provide caregivers with customized supports. By doing so, the students will gain precious experience before they enter the workforce. This proposal will develop and test the effectiveness of this collaborative model. This study will use a randomized controlled design with about a 4- month intervention period. The assessments will take place at baseline, 2 months and 4 months. The study period will be two years. Participants will be 60 convenience family caregivers of the PACE enrollees in Western New York; therefore, CRs are 55 years old or older, need a nursing home level of care, but remain living in the community. Caregivers are adults who visit the CR at least once a week. OTGS will contact the caregivers, using a phone, and conduct an in depth interview to understand their difficulties. Then solutions will be brainstormed amongst OTs and geriatric specialists, and interventions will be formed. At the first visit to the CRs' homes, interviews will be conducted using the Zarit Burden Interview, the Center for Epidemiology Study for Depression, the Buffalo Fatigue Scale, the Positive Aspect of Caregiving, and the Visual Analogue Scale for self-efficacy. The possible solutions will be discussed with caregivers and more detailed difficulties will be videotaped. The solutions that caregivers are comfortable with will be reviewed by the PACE Rehabilitation Department and need to be approved before their implementation. The solutions may include: education of disease process, training for caregivers in supporting CR's activities of daily living (ADL) and instrumental ADL, coordination of family caregivers, problematic behaviors, functional exercise, fall prevention, and increased number of CR's visits to a PACE daycare facility. Statistical analysis will use Generalized Estimating Equations to compare the two groups' linear trends. We expect CRs' condition will deteriorate but the treatment group will reduce caregiver burden and increase self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* • Caregivers of community-dwelling older adults (55 and over) who are member of the PACE

  * Adult 21 years or older
  * Living with the care recipient or within a distance so that they can visit him/her minimum once a week
  * Cognitively intact (can recall three words immediately and 3 minutes later)
  * Competent in English

Exclusion Criteria:

* One instrument (Positive aspect of caregiving) is only available in English. To fully understand caregivers' challenges and convey solutions, our current study OT graduate students are not competent enough in other languages to provide interventions. We do not have budget to hire interpreters.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in caregiver burden measured by the Zarit Burden Interview | 4 months
  To measure changes in burden of care using the 22-item Zarit Burden Interview (ZBI). Each item is rated from Never (0), Rarely (1), Sometimes (2), Quite Frequently (3), to Nearly Always (4). Higher scores indicate higher burden. The ZBI is scored by adding up the responses of all items, ranging from 0 to 88. The interpretations of scores are: 0-20 (no burden), 21-40 (mild to moderate burden), 41-60 (moderate to severe burden), and 61-88 (severe burden). The ZBI has good internal consistency reliability and good validity, and scores were significantly positively correlated with behavior problems in the care recipients and depression scores of the caregivers, according to the study using caregivers (Herbert et al, 2000).
Change in depression change measured by the Center for Epidemiology Studies-Depression | 4 months
  To measure changes in depression using the Center for Epidemiology Studies -Depression (CES-D). This scale asks how often a respondent experienced symptoms associated with depression within the past week. The scale is scored from 0 to 3, with 0 representing rarely or none of the time (less than one day), 1 representing some or a little of the time (1 to 2 days), 2 representing occasionally or a moderate amount of time (3 to 4 days), or 3 representing most or all of the time (5 to 7 days). Total scores could range from 0 (the lowest depression score) to 60 (the highest). A score of 16 or higher indicates a depressive symptom. The CES-D has high internal consistency (Cronbach's alpha =.90) (Cosco et al., 2017), and moderate test-retest reliability (the strongest occurring whiten one to three weeks of time), as well as good measurement validity (Gonzalez et al, 2016).
Change in confidence to continue caring for the care recipient in the future (6 months) | 4 months
  To measure changes in confidence to confine caring for the care recipient using Visual Analogue Scale. It asks caregivers to rate their confidence on a scale of 1 to 10 on Visual Analogue Scale. This assessment asked the caregivers to rate themselves regarding their confidence in in caring for the care recipient in six months. A score of 1 represents no confidence, 5, mid-level confidence, and 10 represents completely confidence.

SECONDARY OUTCOMES:
Change in a cognitive level of care recipients measured by the Global Deterioration Scale | 4 months
  To measure changes in cognition using the Global Deterioration Scale (GDS). The GDS consists of levels 1 to 7. Level 1 indicates "no cognitive decline," Level 2, "very mild cognitive decline/ age associated memory impairment," Level 3, "mild cognitive decline," Level 4,"moderate cognitive decline," Level 5, "moderate dementia," Level 6, "moderately severe dementia," and Level 7, "severe dementia." Therefore, higher scores indicate lower cognition. The GDS has established concurrent validity when compared to the Mini-Mental State Exam with high correlation (Reisberg et al, 1994). It also demonstrated satisfactory clinical/biological validity, compared to CT scan measurements (r= 0.50 for sulcal enlargement scans and r= 0.60 for ventricular dilation scans) and cerebral blood flow (r= 0.70-0.80) (Herndon, 2006). The GDS also has high interrater reliability, ranging in various studies from 0.87 to 0.97 (Herndon, 2006).
Change in instrumental activities of daily living (IADL) of care recipients measured by IADL from the Older Americans Resources and Services | 4 months
  To measure changes in IADL using questionnaires in the Older Americans Resources and Services (OARS) Multidimensional Functional Assessment. The IADL has seven items: using a phone, getting to places out of walking distance, shopping for groceries or clothes, preparing own meals, doing housework, taking medication, and handling money. Each item is rated from 0 to 2: Score 0 indicates "completely unable to do the activity", 1," can do the activity with some help" and 2, "can do the activity without help". The total score ranges between 0 and 14 and higher scores indicate higher function. Intraclass Correlations (ICC) intrarater reliability for was .99 for a short interval (7-10 days) and a long interval (4-6 weeks), and the interrater reliability for a short interval was .98 and for a long interval, .91 (Ottenbacher et al., 1994).

CONTACTS AND LOCATIONS:
Overall Officials: Machiko R Tomita, Ph.D., Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Seeher K, Low LF, Reppermund S, Brodaty H. Predictors and outcomes for caregivers of people with mild cognitive impairment: a systematic literature review. Alzheimers Dement. 2013 May;9(3):346-55. doi: 10.1016/j.jalz.2012.01.012. Epub 2012 Nov 2. PMID 23123229
- [Background] Ottenbacher KJ, Mann WC, Granger CV, Tomita M, Hurren D, Charvat B. Inter-rater agreement and stability of functional assessment in the community-based elderly. Arch Phys Med Rehabil. 1994 Dec;75(12):1297-301. PMID 7993167
- [Background] Gonzalez P, Nunez A, Merz E, Brintz C, Weitzman O, Navas EL, Camacho A, Buelna C, Penedo FJ, Wassertheil-Smoller S, Perreira K, Isasi CR, Choca J, Talavera GA, Gallo LC. Measurement properties of the Center for Epidemiologic Studies Depression Scale (CES-D 10): Findings from HCHS/SOL. Psychol Assess. 2017 Apr;29(4):372-381. doi: 10.1037/pas0000330. Epub 2016 Jun 13. PMID 27295022
- [Background] Reisberg B, Sclan SG, Franssen E, Kluger A, Ferris S. Dementia staging in chronic care populations. Alzheimer Dis Assoc Disord. 1994;8 Suppl 1:S188-205. No abstract available. PMID 8068258
- [Result] Etters L, Goodall D, Harrison BE. Caregiver burden among dementia patient caregivers: a review of the literature. J Am Acad Nurse Pract. 2008 Aug;20(8):423-8. doi: 10.1111/j.1745-7599.2008.00342.x. PMID 18786017
- [Result] Dean K, Wilcock G. Living with mild cognitive impairment: the patient's and carer's experience. Int Psychogeriatr. 2012 Jun;24(6):871-81. doi: 10.1017/S104161021100264X. Epub 2012 Jan 17. PMID 22251799
- [Result] Austrom MG, Lu Y. Long term caregiving: helping families of persons with mild cognitive impairment cope. Curr Alzheimer Res. 2009 Aug;6(4):392-8. doi: 10.2174/156720509788929291. PMID 19689239
- [Result] Beinart N, Weinman J, Wade D, Brady R. Caregiver burden and psychoeducational interventions in Alzheimer's disease: a review. Dement Geriatr Cogn Dis Extra. 2012 Jan;2(1):638-48. doi: 10.1159/000345777. Epub 2012 Dec 15. PMID 23341829
- [Result] Pinquart M, Sorensen S. Correlates of physical health of informal caregivers: a meta-analysis. J Gerontol B Psychol Sci Soc Sci. 2007 Mar;62(2):P126-37. doi: 10.1093/geronb/62.2.p126. PMID 17379673
- See also: Identified current evidence of factors influencing dementia-related caregiver burden — http://www.ncbi.nlm.nih.gov/pubmed/18786017
- See also: MCI results in significant challenges for both patients and their carers. Further work is required in order to establish the best way to help patients and carers meet these challenges — http://www.ncbi.nlm.nih.gov/pubmed/22251799
- See also: Describe common psychological and caregiving issues that can cause stress in family members of persons with mild cognitive impairment (PwMCI) in order to assist family members in providing care and support to the PwMCI while also caring for themselves ov — https://www.ncbi.nlm.nih.gov/pubmed/19689239
- See also: Interventions that are individually tailored to the caregiver are particularly effective at reducing caregiver burden and should be further investigated — https://www.ncbi.nlm.nih.gov/pubmed/23341829
- See also: negative effects of caregiving on physical health are most likely to be found in psychologically distressed caregivers facing dementia-related stressors. — https://www.ncbi.nlm.nih.gov/pubmed/17379673
- See also: Depression and psychological comorbidity, although not as pronounced as in dementia caregivers, are common complications in MCI caregivers — https://www.ncbi.nlm.nih.gov/pubmed/23123229
- See also: Reliability and Validity of the Center for Epidemiologic Studies Depression Scale in a Population-Based Cohort of Middle-Aged U.S. Adults — http://connect.springerpub.com/content/sgrjnm/25/3/476

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT04787068/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT04787068/ICF_001.pdf